CLINICAL TRIAL: NCT05423444
Title: Neural Connectivity Before and After Each of the Three Treatment Phases of Trauma-focused Therapy for Adolescent Posttraumatic Stress
Brief Title: Neural Connectivity During Therapy for Adolescent PTSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Amy Garrett, PhD, Associate Professor, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: HSC20220498H; R01MH127216 (NIH)
Record Dates: First submitted 2022-06-10; First posted 2022-06-21 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: PTSD; Adolescent; Psychological Trauma
Keywords: neuroimaging; psychotherapy; trauma; adolescent
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Psychological Trauma; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial of Trauma-focused Cognitive Behavioral Therapy (TF-CBT) versus Treatment as Usual (TAU)
Who Masked: Participant, Outcomes Assessor
Masking Description: An independent assessor will conduct interviews to quantify symptom severity during and after treatment. The participant will not be given specific information about treatment assignment or the differences between the two treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trauma-focused cognitive behavioral therapy (TF-CBT) (Experimental): Trauma-focused Cognitive Behavioral Therapy (TF-CBT) is an evidence-based psychotherapy that is considered the gold-standard treatment for trauma in youth. The TF-CBT model is flexible but it follows a specific order of phases and components, including psychoeducation, emotion regulation skills, processing the trauma narrative, and safety planning. Sessions are provided weekly for 18-weeks.
  Interventions: Behavioral: TF-CBT
- Treatment As Usual (TAU) (Active Comparator): Treatment as usual (TAU) consists of the standard-of-care psychotherapy as provided by licensed clinicians at a local clinic. The order and choice of techniques is based on the knowledge and preferences of the clinicians. Sessions are provided weekly for 18-weeks.
  Interventions: Behavioral: TAU

INTERVENTIONS:
Behavioral: TF-CBT — evidence-based psychotherapy for trauma in youth
  Arms: Trauma-focused cognitive behavioral therapy (TF-CBT)
Behavioral: TAU — treatment as usual
  Arms: Treatment As Usual (TAU)

SUMMARY:
Posttraumatic stress disorder in adolescence impairs neurobiological networks underlying cognitive, social and emotional skills. Neuroimaging research that seeks to identify the neural mechanisms of treatments for PTSD could lead to novel treatments, but progress has been slow using current methods. The proposed study uses an innovative approach to identify neural mechanisms of specific phases of trauma-focused therapy for youth with PTSD, allowing a new understanding of brain changes associated with the process of therapy.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) during adolescence negatively impacts brain networks underlying cognitive, social, and emotional function. Early intervention is important for mitigating long-term effects, but about 20% of youth do not improve sufficiently with current approaches. By identifying the neurobiological mechanisms of effective therapies, the investigators facilitate the development of novel or personalized treatment approaches for youth with PTSD. However, there has been limited progress in identifying the neural mechanisms of treatment using neuroimaging, partly because most studies collect neuroimaging data at only baseline and end-of-treatment, which collapses across multiple parts of the therapeutic process. The objective of the proposed study is to take a new approach by identifying neural mechanisms associated with specific phases of trauma therapy for youth with PTSD. The central hypothesis is that each phase produces specific brain changes that reflect the acquisition of skills and experiences occurring during that phase. Trauma-Focused Cognitive Behavioral Therapy (TF-CBT) is evidence-based and widely-used to treat children and adolescents with PTSD. It consists of 3 well-defined phases, providing an opportunity to test hypotheses with neuroimaging: changes in executive control networks will occur during the skills phase, changes in limbic networks during the narrative phase, and changes in default mode networks during the consolidation phase. To test these hypotheses, the investigators will recruit N=180 girls and boys, ages 12-17, who have PTSD following interpersonal trauma, such as physical abuse, sexual abuse, or witnessing violence. A randomized controlled trial design will be used to assign participants to either Trauma-focused Cognitive Behavioral Therapy (TF-CBT; provided by study team clinicians who meet fidelity standards) or Treatment as Usual (TAU; provided in the community and does not follow a phased structure). Functional magnetic resonance imaging (fMRI) data will be collected before and after each of the 3 phases of TF-CBT or the same time intervals of TAU. Individual differences in age, sex, dissociative subtype, symptom severity and other variables will be investigated as covariates of phase-related neural changes. Analyses will identify the phases of TF-CBT for which brain regions and networks change for the TF-CBT but not the TAU group. The phase(s) that best predict end-of-treatment symptom improvement also will be identified. Exploratory analyses will use neuroanatomical and white matter diffusivity scans to identify co-occurring changes in brain structure. The proposed innovative study will provide novel information on the neurobiological and cognitive mechanisms associated with the process of trauma therapy for youth with PTSD.

ELIGIBILITY:
Inclusion Criteria:

* ages 12-17 and Tanner stage 2 or above
* history of interpersonal trauma
* PTSD symptoms with a rating of '2' or higher on at least one symptom from each of the 4 clusters, using the Clinician-Administered PTSD Scale for Children and Adolescents, and having a duration of at least one month

Exclusion Criteria:

* current or past use of psychiatric medications
* severe suicidal/homicidal ideation
* current hospitalization
* other current psychotherapy or previous treatment with TF-CBT
* history of head injury with loss of consciousness for >5 minutes
* IQ<85
* major medical illness
* MRI contraindications (metal in body; braces on teeth)
* psychosis, bipolar 1, autism, developmental disorder, panic disorder
* first-degree family member with diagnosis of psychosis or bipolar I disorder
* substance dependence within the past 3 months or current drug use that is frequent

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2022-11-29 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Mean intensity within functional connectivity map of intrinsic network | week 0 (baseline)
  functional MRI scans will be used to assess neural connectivity
Mean intensity within functional connectivity map of intrinsic network | week 6
  functional MRI scans will be used to assess neural connectivity
Mean intensity within functional connectivity map of intrinsic network | week 12
  functional MRI scans will be used to assess neural connectivity
Mean intensity within functional connectivity map of intrinsic network | week 18
  functional MRI scans will be used to assess neural connectivity

SECONDARY OUTCOMES:
Clinician Administered PTSD Scale - children and adolescents (CAPS-CA) | Baseline to week 18
  interview to assess for frequency and severity of PTSD symptoms during the past week

CONTACTS AND LOCATIONS:
Overall Officials: Amy Garrett, PhD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- UT Health Department of Psychiatry, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The data sharing plan and reporting of milestones will conform to all preferred NIMH guidelines, as detailed in the NDA Data sharing terms and conditions. Global unique identifiers (GUIDs) will be generated for each study subject. Data will be submitted to NDA every 6 months. We will provide a data submission agreement. The NDA validation tool will be used frequently. The clinical trial protocol also will be submitted as additional information for every collection. Progress reports will include a statement on the progress of data sharing.
  1. Summary of data to be shared:
     neuroimaging, clinical, demographic, phenotypic, neuropsychological
  2. Description of the data dictionaries used to describe the data set:
     Axis 1 diagnoses, CDI, CAPS-CA, fMRI behavior, beta weights, network correlations
  3. Proposed schedule to validate that the data are compliant with the data dictionary:
  Data will be validated on a quarterly basis
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal
URL: http://nda.nih.gov

DOCUMENTS (1):
  • Informed Consent Form (2024-12-02): https://cdn.clinicaltrials.gov/large-docs/44/NCT05423444/ICF_000.pdf